CLINICAL TRIAL: NCT04088162
Title: The Use of Post-operative Negative Pressure Wound Therapy (NPWT) Dressing in the Prevention of Wound Healing Problems and Infectious Complications After Ostomy Reversal Surgery.
Brief Title: The Use of Post-operative NPWT Dressing in the Prevention of Infectious Complications After Ostomy Reversal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michał Pędziwiatr (Other)
Responsible Party: Sponsor-Investigator, Michał Pędziwiatr, Asoc. Prof., Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JagiellonianU-05
Record Dates: First submitted 2019-08-31; First posted 2019-09-12 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2019-09

CONDITIONS: Stoma Ileostomy; Surgical Wound; Negative Pressure Wound Therapy; Postoperative Wound Infection
MeSH Terms: conditions — Surgical Wound; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Dressing (No Intervention): In case of Control group. After Ileostomy closure skin will be closed by 6 to 8 single no absorbable Monosyn 3-0 (Ethicon, Cincinnati, Ohio., USA) sutures, and sterile standard dressing will be placed.
- Postoperative NPWT dressing (Experimental): In case of NPWT group. After Ileostomy closure skin will be closed by 3 or 4 single no absorbable Monosyn 3-0 (Ethicon, Cincinnati, Ohio., USA) sutures. Between them small sponge "tongues" 1x 0,5x2 cm were placed and over whole incision an NANOVA (KCI USA) negative pressure dressing will be placed. In control group first dressing change was made in 48 hours after operation and then every day until suture removal at 7 postoperative day. In NPWT group NANOVA dressing was taken out at 72 hours. 3 steri-streps were placed between sutures and standard sterile dressing was placed. After it dressing was changed every 24 hours until suture removal at 7 postoperative day.
  Interventions: Device: Postoperative Negative Pressure Wound Therapy KCI NANOVA

INTERVENTIONS:
Device: Postoperative Negative Pressure Wound Therapy KCI NANOVA
  Other Names: Postop. NPWT, Postoperative VAC
  Arms: Postoperative NPWT dressing

SUMMARY:
Introduction: Although negative-pressure wound therapy (NPWT) is likely advantageous for wound healing, the efficacy and safety of its prophylactic use remain unclear. We performed a Randomized Control Trial to assess the usefulness of postoperative NPWT in reduction of postoperative wound healing complications and surgical site infections after diverting ileostomy closure, in the group of patients previously operated for colorectal resection due to cancer.

Materials & Methods: Prospective, randomized study will be conducted. Patients with past history of colorectal cancer laparoscopic surgery with protective loop ileostomy scheduled to undergo ileostomy closure with primary wound closure will be randomly divided into groups with or without NPWT. The primary endpoint are incidence of wound related complications (WRC) (wound healing complications witch required surgical intervention other than suture removal or dressing changing). The secondary endpoints are incidences of Surgical Site Infection (SSI) and length of postoperative hospital stay (LOS) and length of complete wound healing (CWH). Cost analysis will also be performed.

In first step of this study between January 2016 and December 2018 we will asses the usefulness of one of the NPWT devices (NANOVA KCI) in prevention of WHC in established group. The second part of the study will be performed in 2 centers between January 2019 and December 2021. In this step we want to compere other NPWT devices in the same application and to confirm single center outcomes .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Previous colorectal resection with the formation of protective ileostomy due to cancer
* Ileostomy closure surgery as an elective procedure.

Exclusion Criteria:

* Emergency or urgent operation
* Active infection
* Other than ileostomy closure or parastomal hernioplasty operation performed.
* Patents who within 1 week after operation will be re-operated or transferred to Intensive Care Unit or other hospital word due to noninfectious complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of wound management complications | 90 days
  Primary endpoint is described as a reduction of wound healing complications (WHC) after protective ostomy closure in a group of patients previously operated for colorectal cancer with protective ileostomy formation. Wound healing complications are described as any condition of wound which required postoperative intervention other than change of dressing or removing of sutures .
Incidence of wound management complications in groups treated with different types of postopNPWT | 90 days
  The primary endpoint is described as a comparison of reduction of wound healing complications (WHC) after protective ostomy closure in a group of patients previously operated for colorectal cancer with protective ileostomy formation between 3 different postopNPWT devices (KCI NANOVA, Smith&Naphiew PICO and Gynadyne XLR 8) . Wound healing complications are described as any condition of wound which required postoperative intervention other than change of dressing or removing of sutures .

SECONDARY OUTCOMES:
Surgical Site Infections (SSI) Incidence | 90 days
  Secondary endpoints is described as incidence of SSI. Incisional SSI diagnosis criteria included an infection that occurred within 30 days after the operation involving the skin, subcutaneous tissue, or deep soft tissue (e.g. fascia and muscle layers) at the incision site, organ or space according to the criteria of CDC and ECDC for diagnosis of SSI
Postoperative Hospital Stay (LOS) | 90 days
  Secondary endpoints is described as postoperative length of hospital stay (LOS)
Complete wound healing (CWH) time | 90 Days
  Secondary endpoints is described as the duration of complete wound healing (CWH). Complete wound healing was defined as complete closure of the wound without any discharge at the outpatient clinic or reported by patient.

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Oddział kliniczny chirurgii ogólnej, endokrynologicznej i onkologii gastroenterologicznej, Poznan, Wielkopolska
  - 2nd Department of General Surgery, Jagiellonian University, Krakow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wierdak M, Pisarska-Adamczyk M, Wysocki M, Major P, Kolodziejska K, Nowakowski M, Vongsurbchart T, Pedziwiatr M. Prophylactic negative-pressure wound therapy after ileostomy reversal for the prevention of wound healing complications in colorectal cancer patients: a randomized controlled trial. Tech Coloproctol. 2021 Feb;25(2):185-193. doi: 10.1007/s10151-020-02372-w. Epub 2020 Nov 7. PMID 33161523